CLINICAL TRIAL: NCT03344237
Title: High-Sensitivity Cardiac Troponin T in Patients Admitted to the Emergency Department With Atrial Fibrillation in the Era of Novel Oral Anticoagulants - Heidelberg Registry of Atrial Fibrillation
Brief Title: hsTnT in Patients Admitted to the ED With Atrial Fibrillation in the Era of NOACs - Heidelberg Registry of Atrial Fibrillation
Acronym: HERA-FIB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr.med. Dr.med.univ. Mehrshad VAFAIE, Cardiologist, University Hospital Heidelberg
Other Study IDs: HERA-FIB
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Heidelberg Registry of Atrial Fibrillation (HERA-FIB) is to collect data on the prevalence and clinical significance of elevated cardiac troponin in a large registry of unselected patients with atrial fibrillation presenting to an emergency department in the era of novel oral anticoagulants (NOACs).

ELIGIBILITY:
Inclusion Criteria:

* documented atrial fibrillation
* availability of at least one hsTnT measurement

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of approximately 5000 consecutive patients with atrial fibrillation presenting to the emergency department of the Heidelberg University Hospital between March 2013 and June 2017
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Vascular and non-vascular death | Follow up after at least 6 months
Nonfatal myocardial infarction | Follow up after at least 6 months
Stroke/systemic embolism | Follow up after at least 6 months

SECONDARY OUTCOMES:
Stroke, systemic embolism, myocardial infarction, vascular death, non-vascular death, composite endpoint of vascular and non-vascular death, nonfatal MI, stroke/systemic embolism | Follow up after at least 6 months

OTHER OUTCOMES:
Major bleeding by definition of International Society on Thrombosis and Haemostasis (ISTH) | Follow up after at least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehrshad Vafaie, Dr.med.Dr.med.univ., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Department of Cardiology, Angiology and Pneumology, Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg, Germany